CLINICAL TRIAL: NCT03072459
Title: A Retrospective Study of the Navio™ Robotic-assisted Surgical System
Brief Title: A Retrospective Study of the Navio Robotic-assisted Surgical System
Acronym: NAVIO
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-NPFS-11
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Results first posted 2022-05-02 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2021-12

CONDITIONS: Surgical Robotics; Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective, multi-center, cohort study with prospective follow-up and comparison to historical control

DETAILED DESCRIPTION:
Subjects who had previously received the Navio robotic-assisted surgical system for unilateral knee replacement (UKR) were assessed to determine the 2-year safety and effectiveness of the Navio system.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old (at the time of surgery) who have undergone Navio System-assisted UKR at least 2 years prior to enrollment. This includes UKR procedures with all Unicondylar Knee cemented implant designs.
2. Subject had a primary diagnosis of unicompartmental, non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, or avascular necrosis, required correction of functional deformity, or required treatment of fractures that were unmanageable using other techniques.

Exclusion Criteria:

1. Subject received the Navio System-assisted UKR on the index joint as a revision for a previously failed UKR.
2. Subject, in the opinion of the Investigator, had advanced osteoarthritis or joint disease at the time of surgery and was better suited for Total Knee Arthroplasty (TKA).
3. Subject, in the opinion of the Investigator, had a neuromuscular disorder that prohibited control of the index joint.
4. Subject, in the opinion of the Investigator, was morbidly obese.
5. Subject, in the opinion of the Investigator, was contraindicated for UKR.
6. Subject (prospective subjects only), in the opinion of the Investigator, has an emotional or neurological condition including mental illness, mental retardation, drug or alcohol abuse.
7. Subject (prospective subjects only) is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred twenty-eight (128) subjects, including 10% inflation to allow for attrition
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beate Hanson, MD, PhD, Study Director — Smith & Nephew, Inc.
Locations (5):
- United States (5):
  - Hedley Orthopedics, Phoenix, Arizona
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Bronson Orthopedic Specialists, Battle Creek, Michigan
  - OrthoNeuro New Albany, New Albany, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Navio Robotic-assisted Surgical System: Subjects who had previously received the Navio™ robotic-assisted surgical system for UKR were assessed to determine the 2-year safety and effectiveness of the Navio™ system.
Period: Overall Study
Arm/Group | Navio Robotic-assisted Surgical System
Started | 128
Completed | 126
Not Completed | 2
Not completed — Device revised/removed | 1
Not completed — Subject not able to return | 1

BASELINE CHARACTERISTICS:
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 39
  ≥ 60 years | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 122
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 128
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: There was one subject with missing height, weight, and BMI information provided from the site, and thus not included in the results.
  centimeters (cm)
    number analyzed (Participants) | 127
    (all) | 172.1 (10.8)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Population: There was one subject with missing height, weight, and BMI information provided from the site, and thus not included in the results.
  kilograms (kg)
    number analyzed (Participants) | 127
    (all) | 89.9 (18.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: There was one subject with missing height, weight, and BMI information provided from the site, and thus not included in the results.
  kg/m^2
    number analyzed (Participants) | 127
    (all) | 30.3 (5.4)
BMI Category [Count of Participants; unit: Participants] — Population: There was one subject with missing height, weight, and BMI information provided from the site, and thus not included in the results.
  Participants
    < 30 kg/m^2: number analyzed (Participants) | 127
    < 30 kg/m^2 | 66
    ≥ 30 kg/m^2: number analyzed (Participants) | 127
    ≥ 30 kg/m^2 | 61
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 7
  Previous smoker | 31
  Never smoked | 74
  Unknown | 16
Surgical Approach [Count of Participants; unit: Participants]
  Medial parapatellar | 89
  Subvastus / Tissue sparing | 18
  Midvastus | 0
  Lateral parapatellar | 3
  Unknown | 0
  Other | 18
Knee System Type [Count of Participants; unit: Participants]
  Missing | 3
  Smith & Nephew | 108
  Other - Non-Smith & Nephew | 17
Unilateral Knee Replacement Type Used [Count of Participants; unit: Participants]
  Medial | 124
  Lateral | 4
Blood Loss Prevention Method [Count of Participants; unit: Participants]
  Tourniquet | 83
  Aquamantus | 0
  Unknown | 45
  Other | 0
Intra-operative Complications [Count of Participants; unit: Participants]
  Yes | 0
  No | 128
Duration of Surgery [Mean (Standard Deviation); unit: hours] | 1.8 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Navio™ System for Revisions at 2+ Years Post-surgical Implantation Survivorship
Description: Analysis of the absence of device revision (overall survivorship) outcomes assessed from Baseline through 120 weeks post-surgical implantation.
Time Frame: Preoperative (Baseline) and 24, 48, 72, 96, and 120 weeks postoperatively
Population: Safety (SAF) population. The SAF population included all subjects who received the study device and were present for follow-up visits at specified time points.
Measure: Number; unit: participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 128
participants
  Number of Knees with Revisions : Week 0 | 0
  Number of Knees with Revisions : Week 24 | 0
  Number of Knees with Revisions : Week 48: number analyzed (Participants) | 127
  Number of Knees with Revisions : Week 48 | 1
  Number of Knees with Revisions : Week 72: number analyzed (Participants) | 127
  Number of Knees with Revisions : Week 72 | 0
  Number of Knees with Revisions : Week 96: number analyzed (Participants) | 110
  Number of Knees with Revisions : Week 96 | 0
  Number of Knees with Revisions : Week 120: number analyzed (Participants) | 69
  Number of Knees with Revisions : Week 120 | 0

2. Secondary Outcome: Evaluation of Efficacy Based on Knee Society Score (KSS) Assessments
Description: Analysis of KSS from preoperatively (Baseline) up to 36 months postoperatively in 6-months increments to evaluate objective observation, patient satisfaction, and function.
  Objective knee indicators: Range 0-100 points; Patient Satisfaction: Range 0-40 points; and Functional Activities: Range 0-100 points.
  Higher scores indicated a better outcome.
Time Frame: Preoperative (Baseline) and 6, 12, 18, 24, 30, and 36 months postoperatively
Population: The KSS questionnaire assessments were self-reported and not all enrolled subjects completed the questionnaires. See detailed number of participants who completed each response question.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 128
score on a scale
  Objective Knee Indicators: Preoperative: number analyzed (Participants) | 116
  Objective Knee Indicators: Preoperative | 48.6 [8 to 92]
  Objective Knee Indicators: 6 Months Postoperative: number analyzed (Participants) | 88
  Objective Knee Indicators: 6 Months Postoperative | 51.6 [4 to 80]
  Objective Knee Indicators: 12 Months Postoperative: number analyzed (Participants) | 51
  Objective Knee Indicators: 12 Months Postoperative | 49.3 [4 to 78]
  Objective Knee Indicators: 18 Months Postoperative: number analyzed (Participants) | 37
  Objective Knee Indicators: 18 Months Postoperative | 49.9 [14 to 72]
  Objective Knee Indicators: 24 Months Postoperative: number analyzed (Participants) | 57
  Objective Knee Indicators: 24 Months Postoperative | 61.9 [14 to 96]
  Objective Knee Indicators: 30 Months Postoperative: number analyzed (Participants) | 52
  Objective Knee Indicators: 30 Months Postoperative | 63.8 [17 to 96]
  Objective Knee Indicators: 36 Months Postoperative: number analyzed (Participants) | 22
  Objective Knee Indicators: 36 Months Postoperative | 60 [11 to 94]
  Patient Satisfaction: Preoperative: number analyzed (Participants) | 45
  Patient Satisfaction: Preoperative | 14.0 [0 to 40]
  Patient Satisfaction: 6 Months Postoperative: number analyzed (Participants) | 15
  Patient Satisfaction: 6 Months Postoperative | 30.0 [18 to 40]
  Patient Satisfaction: 12 Months Postoperative: number analyzed (Participants) | 23
  Patient Satisfaction: 12 Months Postoperative | 32 [18 to 40]
  Patient Satisfaction: 18 Months Postoperative: number analyzed (Participants) | 8
  Patient Satisfaction: 18 Months Postoperative | 32.8 [20 to 40]
  Patient Satisfaction: 24 Months Postoperative: number analyzed (Participants) | 43
  Patient Satisfaction: 24 Months Postoperative | 34.0 [12 to 40]
  Patient Satisfaction: 30 Months Postoperative: number analyzed (Participants) | 34
  Patient Satisfaction: 30 Months Postoperative | 33.4 [18 to 40]
  Patient Satisfaction: 36 Months Postoperative: number analyzed (Participants) | 21
  Patient Satisfaction: 36 Months Postoperative | 34.8 [16 to 40]
  Functional Activities: Preoperative: number analyzed (Participants) | 45
  Functional Activities: Preoperative | 42.8 [0 to 100]
  Functional Activities: 6 Months Postoperative: number analyzed (Participants) | 15
  Functional Activities: 6 Months Postoperative | 73.3 [30 to 98]
  Functional Activities: 12 Months Postoperative: number analyzed (Participants) | 23
  Functional Activities: 12 Months Postoperative | 78.2 [42 to 100]
  Functional Activities: 18 Months Postoperative: number analyzed (Participants) | 8
  Functional Activities: 18 Months Postoperative | 73.9 [43 to 91]
  Functional Activities: 24 Months Postoperative: number analyzed (Participants) | 43
  Functional Activities: 24 Months Postoperative | 81.9 [39 to 100]
  Functional Activities: 30 Months Postoperative: number analyzed (Participants) | 34
  Functional Activities: 30 Months Postoperative | 81.1 [43 to 100]
  Functional Activities: 36 Months Postoperative: number analyzed (Participants) | 21
  Functional Activities: 36 Months Postoperative | 82.6 [55 to 98]

3. Secondary Outcome: Evaluation of Efficacy Based on Veterans RAND 12 (VR-12) Assessments
Description: Analysis of VR-12 scores preoperatively (Baseline) through 36 months postoperatively in 6 months increments. These scores encompass the individual domains of physical component score (PCS), mental component score (MCS) as well as the sub-domain scores within the PCS (physical functioning, role physical, bodily pain, and general health) and those within the MCS (vitality, social functioning, role emotional, and mental health).
  Domain Scores:
  Physical Component Score (PCS): Range 1 to 20 Mental Component Score (MCS): Range 1 to 25
  Sub-domain Scores:
  Physical Functioning: Range 1 to 6 Role Physical: Range 1 to 4 Bodily Pain: Range 1 to 6 General Health: Range 1 to 6 Vitality: Range 1 to 6 Social Functioning: Range 1 to 6 Role Emotional: Range 1 to 4 Mental Health: Range 1 to 10
  Transformation of raw scale scores (range 0-100) = {(actual raw score - lowest possible raw score)/possible raw score range} x100
  A higher score indicates a better outcome.
Time Frame: Preoperative (Baseline) and 6, 12, 18, 24, 30, and 36 months postoperatively
Population: The VR-12 questionnaire assessments were self-reported and not all enrolled subjects completed the questionnaires. See detailed number of participants who completed each response question.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 128
score on a scale
  PCS: Preoperative: number analyzed (Participants) | 44
  PCS: Preoperative | 11.2 [6 to 15]
  PCS: 6 Months Postoperative: number analyzed (Participants) | 25
  PCS: 6 Months Postoperative | 15.0 [11 to 17]
  PCS: 12 Months Postoperative: number analyzed (Participants) | 25
  PCS: 12 Months Postoperative | 15.0 [11.4 to 20]
  PCS: 18 Months Postoperative: number analyzed (Participants) | 9
  PCS: 18 Months Postoperative | 14.9 [12.4 to 17]
  PCS: 24 Months Postoperative: number analyzed (Participants) | 43
  PCS: 24 Months Postoperative | 14.6 [9 to 19]
  PCS: 30 Months Postoperative: number analyzed (Participants) | 36
  PCS: 30 Months Postoperative | 15.0 [11.4 to 17]
  PCS: 36 Months Postoperative: number analyzed (Participants) | 22
  PCS: 36 Months Postoperative | 15.4 [11.4 to 17.4]
  MCS: Preoperative: number analyzed (Participants) | 44
  MCS: Preoperative | 17.3 [10 to 26]
  MCS: 6 Months Postoperative: number analyzed (Participants) | 25
  MCS: 6 Months Postoperative | 19.7 [11 to 26]
  MCS: 12 Months Postoperative: number analyzed (Participants) | 25
  MCS: 12 Months Postoperative | 20.0 [16 to 23]
  MCS: 18 Months Postoperative: number analyzed (Participants) | 9
  MCS: 18 Months Postoperative | 20.1 [18 to 23]
  MCS: 24 Months Postoperative: number analyzed (Participants) | 43
  MCS: 24 Months Postoperative | 20.4 [13 to 24]
  MCS: 30 Months Postoperative: number analyzed (Participants) | 36
  MCS: 30 Months Postoperative | 21.1 [16 to 24]
  MCS: 36 Months Postoperative: number analyzed (Participants) | 22
  MCS: 36 Months Postoperative | 18.6 [2 to 23]

4. Secondary Outcome: Preoperative Evaluation of Efficacy Based on Radiographic Findings
Description: Changes in radiographic findings (anterior-posterior [AP] and lateral x-rays) from Baseline to 3 years postoperatively were collected for the SAF population.
Time Frame: Preoperative (Baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 128
Participants
  Tibial Osteolysis: Yes | 0
  Tibial Osteolysis: No | 0
  Tibial Osteolysis: Unknown | 0
  Tibial Osteolysis: Missing | 128
  Femoral osteolysis: Yes | 0
  Femoral osteolysis: No | 0
  Femoral osteolysis: Unknown | 0
  Femoral osteolysis: Missing | 128
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 0
  Tibial Migration/Subsidence: Unknown | 0
  Tibial Migration/Subsidence: Missing | 128
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 0
  Femoral Migration/Subsidence: Unknown | 0
  Femoral Migration/Subsidence: Missing | 128
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 0
  Heterotropic Ossification: Unknown | 0
  Heterotropic Ossification: Missing | 128
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 0
  Patellar Subluxation: Unknown | 0
  Patellar Subluxation: Missing | 128
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 0
  Patellar Dislocation: Unknown | 0
  Patellar Dislocation: Missing | 128

5. Secondary Outcome: Postoperative 6-Month Evaluation of Efficacy Based on Radiographic Findings
Description: Changes in radiographic findings (AP and lateral x-rays) from Baseline to 3 years postoperatively were collected for the SAF population.
Time Frame: 6 months postoperatively
Population: The data presented for this outcome are based upon the number of participants who returned for evaluation at this specific time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 127
Participants
  Tibial Osteolysis: Yes | 0
  Tibial Osteolysis: No | 25
  Tibial Osteolysis: Unknown | 3
  Tibial Osteolysis: Missing | 99
  Femoral Osteolysis: Yes | 0
  Femoral Osteolysis: No | 25
  Femoral Osteolysis: Unknown | 3
  Femoral Osteolysis: Missing | 99
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 25
  Tibial Migration/Subsidence: Unknown | 3
  Tibial Migration/Subsidence: Missing | 99
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 25
  Femoral Migration/Subsidence: Unknown | 3
  Femoral Migration/Subsidence: Missing | 99
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 25
  Heterotropic Ossification: Unknown | 3
  Heterotropic Ossification: Missing | 99
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 25
  Patellar Subluxation: Unknown | 3
  Patellar Subluxation: Missing | 99
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 25
  Patellar Dislocation: Unknown | 3
  Patellar Dislocation: Missing | 99

6. Secondary Outcome: Postoperative 12-Month Evaluation of Efficacy Based on Radiographic Findings
Description: as for outcome 5
Time Frame: 12 months postoperatively
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 58
Participants
  Tibial Osteolysis: Yes | 1
  Tibial Osteolysis: No | 24
  Tibial Osteolysis: Unknown | 3
  Tibial Osteolysis: Missing | 30
  Femoral Osteolysis: Yes | 0
  Femoral Osteolysis: No | 25
  Femoral Osteolysis: Unknown | 3
  Femoral Osteolysis: Missing | 30
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 25
  Tibial Migration/Subsidence: Unknown | 3
  Tibial Migration/Subsidence: Missing | 30
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 25
  Femoral Migration/Subsidence: Unknown | 3
  Femoral Migration/Subsidence: Missing | 30
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 25
  Heterotropic Ossification: Unknown | 3
  Heterotropic Ossification: Missing | 30
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 25
  Patellar Subluxation: Unknown | 3
  Patellar Subluxation: Missing | 30
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 25
  Patellar Dislocation: Unknown | 3
  Patellar Dislocation: Missing | 30

7. Secondary Outcome: Postoperative 18-Month Evaluation of Efficacy Based on Radiographic Findings
Description: as for outcome 5
Time Frame: 18 months postoperatively
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 41
Participants
  Tibial Osteolysis: Yes | 0
  Tibial Osteolysis: No | 27
  Tibial Osteolysis: Unknown | 0
  Tibial Osteolysis: Missing | 14
  Femoral Osteolysis: Yes | 1
  Femoral Osteolysis: No | 26
  Femoral Osteolysis: Unknown | 0
  Femoral Osteolysis: Missing | 14
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 27
  Tibial Migration/Subsidence: Unknown | 0
  Tibial Migration/Subsidence: Missing | 14
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 27
  Femoral Migration/Subsidence: Unknown | 0
  Femoral Migration/Subsidence: Missing | 14
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 27
  Heterotropic Ossification: Unknown | 0
  Heterotropic Ossification: Missing | 14
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 27
  Patellar Subluxation: Unknown | 0
  Patellar Subluxation: Missing | 14
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 27
  Patellar Dislocation: Unknown | 0
  Patellar Dislocation: Missing | 14

8. Secondary Outcome: Postoperative 24-Month Evaluation of Efficacy Based on Radiographic Findings
Description: as for outcome 5
Time Frame: 24 months postoperatively
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 61
Participants
  Tibial Osteolysis: Yes | 1
  Tibial Osteolysis: No | 22
  Tibial Osteolysis: Unknown | 5
  Tibial Osteolysis: Missing | 33
  Femoral Osteolysis: Yes | 0
  Femoral Osteolysis: No | 24
  Femoral Osteolysis: Unknown | 4
  Femoral Osteolysis: Missing | 33
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 26
  Tibial Migration/Subsidence: Unknown | 2
  Tibial Migration/Subsidence: Missing | 33
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 26
  Femoral Migration/Subsidence: Unknown | 2
  Femoral Migration/Subsidence: Missing | 33
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 26
  Heterotropic Ossification: Unknown | 2
  Heterotropic Ossification: Missing | 33
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 26
  Patellar Subluxation: Unknown | 2
  Patellar Subluxation: Missing | 33
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 26
  Patellar Dislocation: Unknown | 2
  Patellar Dislocation: Missing | 33

9. Secondary Outcome: Postoperative 30-Month Evaluation of Efficacy Based on Radiographic Findings
Description: as for outcome 5
Time Frame: 30 months postoperatively
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 56
Participants
  Tibial Osteolysis: Yes | 0
  Tibial Osteolysis: No | 29
  Tibial Osteolysis: Unknown | 1
  Tibial Osteolysis: Missing | 26
  Femoral Osteolysis: Yes | 0
  Femoral Osteolysis: No | 29
  Femoral Osteolysis: Unknown | 1
  Femoral Osteolysis: Missing | 26
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 30
  Tibial Migration/Subsidence: Unknown | 0
  Tibial Migration/Subsidence: Missing | 26
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 30
  Femoral Migration/Subsidence: Unknown | 0
  Femoral Migration/Subsidence: Missing | 26
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 30
  Heterotropic Ossification: Unknown | 0
  Heterotropic Ossification: Missing | 26
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 30
  Patellar Subluxation: Unknown | 0
  Patellar Subluxation: Missing | 26
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 30
  Patellar Dislocation: Unknown | 0
  Patellar Dislocation: Missing | 26

10. Secondary Outcome: Postoperative 36-Month Evaluation of Efficacy Based on Radiographic Findings
Description: as for outcome 5
Time Frame: 36 months postoperatively
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Navio Robotic-assisted Surgical System
Number analyzed (Participants) | 23
Participants
  Tibial Osteolysis: Yes | 0
  Tibial Osteolysis: No | 13
  Tibial Osteolysis: Unknown | 0
  Tibial Osteolysis: Missing | 10
  Femoral Osteolysis: Yes | 0
  Femoral Osteolysis: No | 13
  Femoral Osteolysis: Unknown | 0
  Femoral Osteolysis: Missing | 10
  Tibial Migration/Subsidence: Yes | 0
  Tibial Migration/Subsidence: No | 13
  Tibial Migration/Subsidence: Unknown | 0
  Tibial Migration/Subsidence: Missing | 10
  Femoral Migration/Subsidence: Yes | 0
  Femoral Migration/Subsidence: No | 13
  Femoral Migration/Subsidence: Unknown | 0
  Femoral Migration/Subsidence: Missing | 10
  Heterotropic Ossification: Yes | 0
  Heterotropic Ossification: No | 13
  Heterotropic Ossification: Unknown | 0
  Heterotropic Ossification: Missing | 10
  Patellar Subluxation: Yes | 0
  Patellar Subluxation: No | 13
  Patellar Subluxation: Unknown | 0
  Patellar Subluxation: Missing | 10
  Patellar Dislocation: Yes | 0
  Patellar Dislocation: No | 13
  Patellar Dislocation: Unknown | 0
  Patellar Dislocation: Missing | 10

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from Study Day 1 until up to 2 years postoperatively (+/- 3 months) at End of Study.
Arm/Group | Navio Robotic-assisted Surgical System
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 2/128
Other Adverse Events (participants affected / at risk) | 28/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navio Robotic-assisted Surgical System (N=128)
Deep venous thrombosis (DVT) (Vascular disorders) | 1 (1) — The subject recovered/resolved from the DVT and it was deemed unrelated to the treatment. The subject was not discontinued from the study.
Lower extremity DVT (Vascular disorders) | 1 (1) — The subject recovered/resolved from the DVT and it was deemed unrelated to the treatment. The subject was not discontinued from the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navio Robotic-assisted Surgical System (N=128)
Radiolucency line tibial ML zone (Musculoskeletal and connective tissue disorders) | 5 (5)
Redness, burning, itchiness (Skin and subcutaneous tissue disorders) | 1 (1)
Effusion (Skin and subcutaneous tissue disorders) | 1 (1)
Swelling and discomfort (Skin and subcutaneous tissue disorders) | 1 (1)
Slight swelling and edema (Skin and subcutaneous tissue disorders) | 1 (1)
Knee pain due to mild iliotibial band tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in quadriceps (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain with 50 mL of blood aspiration (Musculoskeletal and connective tissue disorders) | 1 (1)
Possible cellulitis - not life threatening (Skin and subcutaneous tissue disorders) | 1 (1)
Manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 1 (1)
Occasional swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Soreness/pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Incisional soreness (Skin and subcutaneous tissue disorders) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pin site drainage (Skin and subcutaneous tissue disorders) | 1 (1)
Pimple drainage from pin site (Skin and subcutaneous tissue disorders) | 1 (1)
Stress shielding (Musculoskeletal and connective tissue disorders) | 1 (1)
Radiolucent lines (Musculoskeletal and connective tissue disorders) | 7 (7)
Femoral osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Incision pain with deep flexion (Skin and subcutaneous tissue disorders) | 1 (1)
Anterior knee pain and swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial hypertrophy, quadriceps atrophy, and knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hamstring irritation and ischial tuberosity bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin irritation over pin site (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no known study limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT03072459/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT03072459/SAP_001.pdf